CLINICAL TRIAL: NCT00756873
Title: Analgesic Efficacy and Safety of Etoricoxib in Ear Nose Throat Surgery
Brief Title: Etoricoxib in Ear Nose Throat Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Regensburg (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Michael Bucher, MD, PhD, University Hospital Regensburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Etoric-TE-1
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Tonsillectomy
Keywords: Elective tonsillectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: Administration of placebo
- 2 (Experimental): Etoricoxib 90 mg qd.
  Interventions: Drug: Administration of etoricoxib
- 3 (Experimental): Etoricoxib 120 mg qd. (day 0-7) Etoricoxib 90 mg qd. (day 8-14)
  Interventions: Drug: Administration of etoricoxib

INTERVENTIONS:
Drug: Administration of placebo — Placebo qd orally day 0-14
  Arms: 1
Drug: Administration of etoricoxib — Etoricoxib 90 mg qd orally day 0-14
  Arms: 2
Drug: Administration of etoricoxib — Etoricoxib 120 mg qd orally day 0-7 Etoricoxib 90 mg qd orally day 8-14
  Arms: 3

SUMMARY:
The aim of this study is to test the analgesic efficacy of etoricoxib (90 mg or 120 mg qd. perioperatively) for post-operative pain relief.

The primary endpoint is as follows:

* does preoperative etoricoxib reduce the post-operative opioid utilization in patients undergoing elective tonsillectomy under general anaesthesia (i.e. the post-operative opioid-sparing effect of etoricoxib in humans).

The secondary endpoints are as follows:

* does the etoricoxib medication have an impact on PONV or activities of daily
* does the etoricoxib medication influence the blood loss during surgery or the incidence of postoperative bleeding
* does the etoricoxib medication influence the operation time. In addition, adverse effects of etoricoxib will be documented.

DETAILED DESCRIPTION:
On day of surgery (day 0) the patients will be randomly assigned to one of the three groups using a sealed envelope method. The etoricoxib 90 mg group receives etoricoxib (Arcoxia®, Merck Sharp & Dohme GmbH, Haar, Germany) 90 mg orally, the etoricoxib 120 mg group receives etoricoxib 120 mg orally and the control group receives a placebo tablet orally 1 h before surgery (day 0). All patients receive a standard general anesthesia with intravenous propofol (2-3 mg/kg), fentanyl (2 µg/kg) and mivacurium (0.2 mg/kg) for induction. Patients are ventilated via a tracheal tube, anesthesia being maintained with sevoflurane (0.8 - 1.5% end-tidal concentration). If mean arterial blood pressure or heart rate increase to more than 25% above the pre-operative baseline value despite an end-tidal concentration of 1.5% sevoflurane, an intravenous bolus of fentanyl 0.05 mg will be administered. Monitoring includes electrocardiogram (ECG), non-invasive arterial blood pressure, pulse oximetry, end-tidal CO2 and end-tidal sevoflurane. On days 1 to 3 patients will receive etoricoxib (90 mg or 120 mg qd.) or placebo. After discharge on day 3, patients will receive etoricoxib (90 mg or 120 mg qd.) or placebo until cessation of pain during activity (swallowing). According to the current label for Arcoxia® 120 mg in Germany, patients taking etoricoxib 120 mg will switch to etoricoxib 90 mg on day 8. Rescue medication will be piritramid i.v. (day 0), oxycodone p.o. (day 1-2) and paracetamol p.o. (day 3-14).

Day -7 to -1: Inclusion/exclusion criteria, medical history, concomitant medications, laboratory, serum pregnancy test, informed consent Day 0: Study medication 1 h before surgery, intra-operative blood loss, pain score, opioid utilization, PONV score and anti-emetic medication Day 1: pain score, opioid utilization, PONV score, anti-emetic medication, bleeding Day 2: pain score, opioid utilization, PONV score, anti-emetic medication, bleeding Day 3: pain score, opioid utilization, PONV score, anti-emetic medication, bleeding Day 7: pain score, paracetamol utilization, bleeding Day 14: first day with no pain, last study medication, paracetamol utilization, bleeding

ELIGIBILITY:
Inclusion Criteria:

* male or female patients
* 18 years of age
* female patients not pregnant/non-lactating
* indication for elective tonsillectomy
* written informed consent.

Exclusion Criteria:

* etoricoxib, other analgesic or anti-emetic medication within 10 half-lives
* evidence for active peptic ulceration
* history of gastrointestinal bleeding
* evidence of hepatic, renal or hematopoietic disorders
* heart failure (NYHA II-IV)
* uncontrolled arterial hypertension
* clinical evidence of arterial occlusive disease
* coronary heart disease or cerebrovascular disease
* inflammatory bowel disease
* hypersensitivity to analgetics, antipyretics, NSAIDs or antiemetics
* evidence for noncompliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-09 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative opioid-sparing effect of etoricoxib in humans undergoing elective tonsillectomy | Day 0-3 after surgery

SECONDARY OUTCOMES:
Impact of etoricoxib medication on PONV or activities of daily or the incidence of postoperative bleeding | Day 0-14

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Universtiy Hospital Regensburg, Regensburg
  - Weiden Clinic, Weiden I.d. OPf.